CLINICAL TRIAL: NCT04893499
Title: The Effectiveness of a Natural Aqueous Extract of Chios Mastic in the Management of Irritable Bowel Syndrome: the MASTIQUA Randomized Controlled Clinical Trial
Brief Title: A Study of Chios Mastic Water in Irritable Bowel Syndrome
Acronym: MASTIQUA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Harokopio University (Other)
Responsible Party: Principal Investigator, Labros Sidossis, Ph.D., Professor in Nutrition - Dietetics, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Γ-1038/12-3-2021
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Pistacia Lentiscus var. Chia; Chios mastic; mastiha; irritable bowel syndrome; dyspepsia; constipation; diarrhea; abdominal pain; bloating; gastrointestinal health
MeSH Terms: conditions — Irritable Bowel Syndrome; Dyspepsia; Constipation; Diarrhea; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-dose mastic group (Experimental): This arm will consume 600 mL of a sparkling water enriched with Chios mastic per day for a 3-month period.
  Interventions: Behavioral: Chios mastic water
- Low-dose control group (Placebo Comparator): This arm will consume 600 mL of a standard sparkling water per day for a 3-month period.
  Interventions: Behavioral: Placebo water
- High-dose mastic group (Experimental): This arm will consume 600 mL of a sparkling fruit juice enriched with Chios mastic per day for a 3-month period.
  Interventions: Behavioral: Chios mastic fruit juice
- High-dose control group (Placebo Comparator): This arm will consume 600 mL of a standard sparkling fruit juice per day for a 3-month period.
  Interventions: Behavioral: Placebo fruit juice

INTERVENTIONS:
Behavioral: Chios mastic water — Participants randomized to this intervention arm will be provided with a sparkling water enriched with the natural mastic aqueous extract (0.06%), a by-product of Chios mastic processing, and will be asked to consume it daily (3 bottles of 200 mL each) for 3 months. Participants will also be instructed to keep the use of medication and dietary supplements stable and preserve their typical lifestyle habits throughout the study.
  Other Names: Mastiqua
  Arms: Low-dose mastic group
Behavioral: Placebo water — Participants randomized to this intervention arm will be provided with a standard sparkling water and will be asked to consume it daily (3 bottles of 200 mL each) for 3 months. Participants will also be instructed to keep the use of medication and dietary supplements stable and preserve their typical lifestyle habits throughout the study.
  Arms: Low-dose control group
Behavioral: Chios mastic fruit juice — Participants randomized to this intervention arm will be provided with a sparkling fruit juice enriched with the natural mastic aqueous extract (0.55%), a by-product of Chios mastic processing, and will be asked to consume it daily (3 bottles of 200 mL each) for 3 months. Participants will also be instructed to keep the use of medication and dietary supplements stable and preserve their typical lifestyle habits throughout the study.
  Other Names: Mastiqua lemon
  Arms: High-dose mastic group
Behavioral: Placebo fruit juice — Participants randomized to this intervention arm will be provided with a standard sparkling fruit juice and will be asked to consume it daily (3 bottles of 200 mL each) for 3 months. Participants will also be instructed to keep the use of medication and dietary supplements stable and preserve their typical lifestyle habits throughout the study.
  Arms: High-dose control group

SUMMARY:
Chios mastic is a natural product with strong antimicrobial, anti-inflammatory and antioxidant properties, and well-established benefits for dyspeptic disorders. The aim of the present study is to investigate the effectiveness of a natural aqueous extract of Chios mastic (mastic water), a by-product of Chios mastic processing, in the management of irritable bowel syndrome. This will be a 3-month randomized double-blind controlled clinical trial in adult patients with irritable bowel syndrome under standard medication. Participants will be blindly randomized to a low-dose mastic group, which will receive a carbonated water enriched with Chios mastic water (0.06%), a high-dose mastic group, which will receive a carbonated fruit juice enriched with Chios mastic water (0.55%), or one of the two control groups, which will receive an identical placebo water/fruit juice with no active ingredients. Participants will be evaluated in terms of anthropometric indices, lifestyle habits, severity of IBS-related gastrointestinal symptoms, quality of life, as well as biochemical, inflammatory and oxidative stress markers, both pre- and post-intervention.

DETAILED DESCRIPTION:
Chios mastic is the resin of the mastic tree (Pistacia Lentiscus var. Chia), produced exclusively in the southern part of the Greek island of Chios. References about its medical use from local populations for the treatment of gastrointestinal disorders or as a cosmetic agent can be found in ancient texts. Nowadays, this versatile resin has been rediscovered, not only as a traditional remedy and aromatic agent, but as a potent phytotherapeutic product with strong anti-inflammatory, anti-microbial and anti-oxidant properties. In 2015, Chios mastic was recognized as a herbal medicinal product by the European Medicines Agency (EMA), with two therapeutic indications: mild dyspeptic disorders and skin inflammation/healing of minor wounds (EMA/HMPC/46758/2015). Over the last years, Chios mastic is widely used in medicinal products, food supplements and cosmetics and has become the object of intense study in the fields of Nutrition and Pharmacotechnology.

Irritable bowel syndrome (IBS) is a chronic functional gastrointestinal disease characterized by adverse changes in bowel function (frequency of bowel movements and/or stool composition) and abdominal pain. The clinical presentation of IBS usually includes symptoms of abdominal pain, flatulence, bloating, diarrhea and constipation that often alternate, while postprandial discomfort in the upper abdomen, feeling of fullness, nausea, vomiting and back pain are less commonly reported. IBS affects approximately 7-16% of the general population, and leads to reduced functionality and productivity and a significant deterioration in quality of life due to its various intestinal manifestations. The first-line pharmacological treatments for IBS aim at alleviating symptoms and include antispasmodics or anticonvulsants for abdominal pain, antidiarrheal medication and laxatives for constipation. Dietary modifications, such as the avoidance of foods that aggravate gastrointestinal symptoms and various types of exclusion diets, are also applied as adjunctive therapies for IBS management, but evidence of their effectiveness remains scares and inconclusive.

The use of foods/beverages enriched with Chios mastic could constitute a promising complementary approach for the management of IBS, in combination with current first-line pharmacological treatments. The aim of the present interventional study is to explore the effectiveness of a natural aqueous extract of Chios mastic in the management of IBS.

The study will be a 3-month parallel, randomized (allocation ratio 1:1), controlled, double-blind clinical trial in a sample of 60 adult patients with IBS. Eligible participants will be adult (18-65 years old) otherwise healthy individuals with an IBS diagnosis based on ROME IV criteria under stable medication. Participants will be excluded on the basis of the presence of other chronic gastrointestinal diseases, the presence of other serious comorbidities, or recent significant changes in lifestyle habits. Participants will be randomized to a low-dose mastic group (LDMG), a low-dose control group (LDCC), a high-dose mastic group (HDMG) or a high-dose control group (HDCC). The LDMG will be provided with 600 mL of a sparkling water (mastiqua) containing the natural mastic aqueous extract (0.06%) to be consumed daily (3 bottles of 200 mL each). The HDMG will be provided with 600 mL of a sparkling fruit juice (mastiqua lemon) containing the natural mastic aqueous extract (0.55%) to be consumed daily (3 bottles of 200 mL each). The LDCC and HDCC will receive the same quantity of a placebo sparkling water or fruit juice, respectively. For each type of drink (water and fruit juice), the intervention and placebo drinks will be unlabeled and identical in appearance and organoleptic characteristics, including the characteristic Chios mastic aroma. Randomization will be performed by an investigator with no clinical involvement, while all patients and study team members will be blinded to patient allocation in study groups.

All enrolled patients will continue their standard medical treatment which must remain stable throughout the trial. The study physician will systematically record potential side-effects and will be in charge of terminating the intervention if needed. Participants will be assessed in terms of anthropometric indices (body weight, height, waist circumference, and body composition), lifestyle habits (diet and physical activity habits), the presence and severity of gastrointestinal symptoms, and quality of life both pre- and post-intervention. In addition, blood samples after a 12-hour fast and morning urine samples will be collected to measure biochemical, inflammatory and oxidative stress markers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Body mass index 18.5-35 kg/m2
3. IBS diagnosis

Exclusion Criteria:

1. Presence of other gastrointestinal disorders, such as gastritis, peptic ulcer, functional dyspepsia, celiac disease and inflammatory bowel disease
2. Presence of other serious comorbidities, such as diabetes mellitus, active cancer, cardiovascular disease, pulmonary, kidney, liver, chronic inflammatory, autoimmune or psychiatric diseases
3. Recent (within 6 months) surgery or hospitalization
4. Habitual excessive alcohol consumption (> 210 or > 140 gr of alcohol per week for men and women, respectively)
5. Currently on a weight-loss diet or recent change (within 6 months) in lifestyle habits
6. Pregnancy or breast feeding (for women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-09-12 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Change in IBS symptoms severity assessed through the IBS Symptom Severity Scale (IBS-SSS) | 0 (baseline) and 12 weeks
  The score ranges from 0 to 500, with higher values indicating more severe symptoms.
Change in quality of life assessed through the IBS Quality of Life questionnaire (IBS-QOL) | 0 (baseline) and 12 weeks
  Τhe score ranges from 34 to 170 with higher values indicating lower quality of life.

SECONDARY OUTCOMES:
Change in high-sensitivity C-reactive protein | 0 (baseline) and 12 weeks
  High-sensitivity C-reactive protein (mg/L) will be measured in blood samples by nephelometry.
Change in high-sensitivity interleukin-6 levels | 0 (baseline) and 12 weeks
  High-sensitivity interleukin-6 levels (pg/mL) will be measured in blood samples using commercially available ELISA kits.
Change in malondialdehyde | 0 (baseline) and 12 weeks
  Malondialdehyde levels (nmol/mL) will be measured in blood samples through HPLC-Fluorescence.
Change in total serum antioxidant capacity | 0 (baseline) and 12 weeks
  Total serum antioxidant capacity (μmol/L) will be measured in blood samples using commercially available ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Labros Sidossis, PhD, Principal Investigator — Department of Kinesiology and Health, School of Arts and Sciences, Rutgers University; Michael Georgoulis, PhD, Study Chair — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University; Alexandra Karachaliou, MSc, Study Chair — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University
Locations (1):
- Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared to investigators for the purpose of data meta-analysis, provided that the proposed use of the data has been approved by the Study Principal Investigator. Proposals should be directed to lsidossis@gmail.com. To gain access, data requestors will need to sign a data access agreement.